CLINICAL TRIAL: NCT00740675
Title: Ambulatory Medication Reconciliation Following Hospital Discharge: Project 4 From "Center for Education and Research on Therapeutics (CERT) on Health Information Technology"
Brief Title: Ambulatory Medication Reconciliation Following Hospital Discharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Jeffrey L. Schnipper, MD, MPH, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1U18 HS016790-01
Record Dates: First submitted 2007-12-28; First posted 2008-08-25 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Medication Administered in Error; Adverse Drug Events
Keywords: adverse drug events; outpatient
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): At post-discharge follow-up visit with PCP, PCP views:
  1. Discharge medication reconciliation screen.
  2. Prompts to perform post-discharge reconciliation at the first post-discharge visit.
  Interventions: Other: Outpatient Medication Reconciliation
- Uusual care (No Intervention): PCPs manage the patient's medications after hospital discharge as they normally would.

INTERVENTIONS:
Other: Outpatient Medication Reconciliation — The post-discharge medication reconciliation module has the following features:
  1. Presents the (preadmission) ambulatory medication list and the hospital discharge medication list side-by-side, sorted by class, with all identical medications lined up next to each other and all differences in the two regimens highlighted.
  2. Allows users to update the ambulatory medication list with a few keystrokes (i.e., to accept individual changes made during the hospitalization).
  3. Allows reconciliation to be performed in full (e.g., for PCPs who are responsible for the entire medication list) or in part (e.g., for specialists).
  Arms: 1

SUMMARY:
Adverse drug events (ADEs) after hospital discharge are common. The purpose of this research study is see if we can design an electronic tool given to your primary care provider (PCP) that will reduce adverse drug events, hospital readmissions, and emergency department visits after you are discharged from the hospital.

DETAILED DESCRIPTION:
The objective of this research is to reduce the incidence of post-discharge medication discrepancies, preventable and ameliorable ADEs, hospital readmissions, and ED visits through the use of HIT. The proposed tool will prompt primary care physicians to perform medication reconciliation at the first post-discharge outpatient visit, clearly display and organize preadmission and discharge medication regimens, and facilitate the creation of the new post-discharge medication list with just a few keystrokes. Using methodologies from prior studies at BWH, we will evaluate the intervention in a two-site RCT. The study will be conducted at Brigham and Women's Hospital and Massachusetts General Hospital, taking advantage of our rich experience with designing and testing new informatics applications, including one for inpatient medication reconciliation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to BWH or MGH who plan to follow up with a PCP in one of 12 primary care practices affiliated with BWH or MGH.
* Patients will need to meet the following criteria:

  * 1) be 55 years or older,
  * 2) be admitted to the participating delivery system's hospital during the study period for a non-psychiatric condition,
  * 3) have no plans to enter hospice,
  * 4) be discharged back to the community,
  * 5) be prescribed 5 or more medications at discharge, including at least one of the following:

    * antibiotics,
    * insulin,
    * antihypertensives,
    * anti-rejection,
    * antiarrhythmics,
    * inhalers,
    * antiepileptics,
    * antianginals,
    * pain medications,
    * oral hypoglycemics,
    * steroids,
    * anticoagulants.
  * These drugs were selected because they require close monitoring, increase risk for drug-drug interactions, have a narrow therapeutic window, or are known to increase risk for ADEs in the older adult population

Exclusion Criteria:

Unable to provide informed consent and has no proxy who administers patient's medications and can provide informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
presence of at least one serious medication error per patient | 30 days post-discharge

SECONDARY OUTCOMES:
ED visits and non-scheduled hospital readmissions and ED visits | within 30 days of discharge
Accuracy of medication list in ambulatory electronic medical record | 30 days post discharge

CONTACTS AND LOCATIONS:
Overall Officials: David W Bates, MD, MSc, Study Director — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts